CLINICAL TRIAL: NCT06620900
Title: Expanding Access to mTBI Treatment for Veterans and Service Members With Co-occurring Substance Use
Acronym: ExpandAccess
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shepherd Center, Atlanta GA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2156344; TP230246 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Concussion, Mild Traumatic Brain Injury; Brain Injury; Traumatic Brain Injury; Substance Use; Substance Use Disorder (SUD)
Keywords: Concussion; Mild Traumatic Brain Injuty; Brain Injury; Substance use; Substance Use Disorder; Military; Service Members; Veterance; Interdisciplinary; Intensive Outpatient Program; Neurorehabilitation
MeSH Terms: conditions — Brain Concussion; Brain Injuries; Brain Injuries, Traumatic; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Integrated Model of Care (Experimental): Participants will engage in interdisciplinary intensive outpatient program (IOP) treatment for mild traumatic brain injury with individualized support for substance use (SU) following which they will receive support for SU in the transition support program.
  Interventions: Other: Integrated Model of Care

INTERVENTIONS:
Other: Integrated Model of Care — The Integrated Model of Care was developed and piloted by the study team provide support for individuals seeking care in an interdisciplinary intensive outpatient program for mild traumatic brain injury to receive support for co-occurring substance use-related needs.

SUMMARY:
The purpose of this research is to determine whether military veterans and service members with mild traumatic brain injury with and without co-occurring substance use can complete and benefit from integrated interdisciplinary care individualized to their symptoms, goals, and needs.

Participants will complete surveys about substance use and other symptoms at the beginning and end of treatment in an intensive outpatient program and 6 months after discharge.

DETAILED DESCRIPTION:
This pragmatic clinical trial will (1) assess treatment retention and treatment outcomes at the completion of interdisciplinary intensive outpatient program (IOP) and at a 6-month follow-up comparing service members and veterans (SM/Vs) with mild traumatic brain injury (mTBI) + substance use (SU) and a TBI -control group; and (2) assess SU-related outcomes at the end of IOP treatment and durability of SU outcomes at 6-months follow-up among SM/Vs with co-occurring SU. Analyses of these key treatment outcomes along with input from lived experience consultants and other key stakeholders, will be used to refine and disseminate a scalable approach to treating individuals with mTBI and co-occurring SU.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* US military service member or veteran
* Diagnosis of mild traumatic brain injury (mTBI) and/or repetitive head impact/blast exposures
* Participating in the SHARE Military Initiative intensive outpatient program

Exclusion Criteria:

* History of brain injury other than mTBI or progressive neurological disorder
* Active psychosis
* Not able to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Neurobehavioral Symptom Inventory (NSI) | Study enrollment, immediately after the intervention, and at 6 months follow-up
  a 22-item, self-report questionnaire used to measure change in symptoms commonly associated with mild traumatic brain injury over time
Short Inventory of Problems- Revised (SIP-R) | Study enrollment, immediately after the intervention, and at 6 months follow-up
  a 17-item self-report inventory used to assess adverse consequences of substance use

SECONDARY OUTCOMES:
Life-Satisfaction Questionnaire -11 (LISAT-11) | Study enrollment, immediately after the intervention, and at 6 months follow-up
  an internationally validated 11-item self-report inventory of satisfaction within important life domains: life as a whole, vocational situation, financial situation, leisure situation, contacts with friends, sexual life, self-care management, family life, partner, physical health, and psychological health
Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | Study enrollment, immediately after the intervention, and at 6 months follow-up
  a 20-item self-report inventory used to assess severity of posttraumatic stress symptoms and monitoring symptom change during and after treatment
Patient Health Questionnaire (PHQ-8) | Study enrollment, immediately after the intervention, and at 6 months follow-up
  an eight item, self-report inventory used to screen for the presence and severity of depression
Generalized Anxiety Disorder Scale (GAD-7) | Study enrollment, immediately after the intervention, and at 6 months follow-up
  a seven item, self-report inventory used to screen for the presence and severity of anxiety
Repeatable Battery for the Assessment of Neuropsychological Status Update (RBANS Update) | Study enrollment and immediately after the intervention
  a multi-item, multi-subtest, clinician administered objective assessment used to measure change over time in neuropsychological status by yielding a Total Score, as well as Immediate Memory, Delayed Memory, Attention, Language, and Visuospatial/ Constructional scores
Sensory Organization Test (SOT) | Study enrollment and immediately after the intervention
  completed as part of quantitative Balance Testing (Bertec) which provides information about postural stability by measuring subject sway on a force platform under different sensory conditions; the SOT is used to evaluate sensory weighting in postural control using a series of conditions of increased difficulty.
Behavior Rating Inventory of Executive Functioning - Adult Version (BRIEF-A) | Study enrollment and immediately after the intervention
  a 75-item self-report inventory of executive functioning in everyday environments that yields a total Global Executive Composite score as well as a Behavioral Regulation Index and Metacognitive Index
Alcohol Use Disorders Identification Test- Concise (AUDIT-C) | Study enrollment and at 6 months follow-up
  a three-item, self-report screening tool used to identify people who with active alcohol use disorders (including alcohol abuse or dependence).
Drug Abuse Screening Test (DAST-10) | Study enrollment and at 6 months follow-up
  a 10-item self-report instrument that yields a quantitative index of the degree of consequences related to drug use
Cannabis Use Disorder Identification Test (CUDIT-R) | Study enrollment and at 6 months follow-up
  an 8-item measure designed for screening for problematic cannabis use and use a brief repeated outcome measure
National Survey on Drug Use and Health (NSDUH)- 30-day use: Alcohol and Substances | Study enrollment, immediately after the intervention, and at 6 months follow-up
  survey of alcohol use (tallying days used and estimating average number of drinks per drinking day) and additional substances used (number of days used)

CONTACTS AND LOCATIONS:
Locations (1):
- Shepherd Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
We will submit de-identified research data into the Federal Interagency TBI Research (FITBIR) Informatics System at the completion of the clinical trial. The following data will be collected and reported the following National Institute of Neurological Disorders and Stroke (NINDS) TBI common data elements (CDE) as part of this process:
  * Demographics and Injury Characteristics
  * Neurobehavioral Symptom Inventory (NSI)
  * Alcohol Use Disorders Identification Test-Concise (AUDIT-C)
  * Patient Health Questionnaire (8 Item) (PHQ-8)
  * Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5)
  * Behavior Rating Inventory of Executive Function - Adult Version (BRIEF-A)
  * Life-Satisfaction Questionnaire -11 (LISAT-11)
  * Sensory Organization Test (SOT)
  * Short Inventory of Problems- Revised (SIP-R)
  * Drug Abuse Screening Test (DAST-10)
  * Cannabis Use Disorder Identification Test (CUDIT-R)
  * National Survey on Drug Use and Health (NSDUH)- 30-day use: Alcohol and Substances
Time Frame: We will complete upload of IPD by Aug 31, 2025.
Access Criteria: Researchers can then file an application with FITBIR, following FITBIR processes and protocols, to request access to the data for research purposes.

REFERENCES:
- [Background] Wallace TD, McCauley KL, Hodge AT, Moran TP, Porter ST, Whaley MC, Gore RK. Use of person-centered goals to direct interdisciplinary care for military service members and Veterans with chronic mTBI and co-occurring psychological conditions. Front Neurol. 2022 Nov 16;13:1015591. doi: 10.3389/fneur.2022.1015591. eCollection 2022. PMID 36523344
- See also: Related Info — https://www.shepherd.org/research/acquired-brain-injury/mtbi-lab

DOCUMENTS (1):
  • Informed Consent Form (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT06620900/ICF_000.pdf